CLINICAL TRIAL: NCT00572806
Title: Evaluation of the Initiation of Insulin Treatment Using Insulin Aspart on Blood Glucose Profile in Type 2 Diabetes Mellitus
Brief Title: Initiation of Insulin Aspart in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1501
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate if using insulin aspart as start therapy will improve the efficacy on daytime blood glucose cycle profile in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 years
* HbA1c greater than 8.0%
* Body Mass Index (BMI) below 40.0 kg/m2
* Inadequate treatment with diet and OADs
* Never received treatment with insulin

Exclusion Criteria:

* Type 1 diabetes
* Known or suspected allergy to investigational product

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-02-05 (Actual); Primary Completion 2004-02-02 (Actual); Study Completion 2004-02-02 (Actual)

PRIMARY OUTCOMES:
Blood glucose value | at 5 pm in a daytime blood glucose cycle profile

SECONDARY OUTCOMES:
Evaluation of 24-hour blood glucose cycle
HbA1c
Hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Montpellier, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com